CLINICAL TRIAL: NCT04466462
Title: Cross-sectional Study of COVID-19 Infection in Hospital Health Personnel
Status: Completed | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-Hosp
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to determine the percentage of past SARS-CoV-2 infections in hospital health personnel involved in the care of people with COVID-19 in HUGTiP and in Badalona Serveis Assistencials de Badalona.

DETAILED DESCRIPTION:
Health personnel, especially hospital workers, have been a group especially affected by the COVID-19 epidemic. According to data from the Ministry of Health, in Spain 26% of health personnel have been infected by COVID-19, for a total of 31,053 professionals, representing up to 18.5% of all infections in the Spanish state, with variations between the different autonomous communities.1 In Italy it was estimated that up to 20% of health workers who responded to the epidemic would have been infected within a month.

There are no unified guidelines at the state level to determine infection prevention strategies in health personnel in order to validate them, beyond the use of Personal Protective Equipment (PPE) in personnel and general strategies for isolation and prevention of transmission.

There are no approved drug prevention strategies for primary prophylaxis against COVID-19.

Currently, there are no universal mass screening strategies (virological or immunological) to estimate the actual number of health personnel with an asymptomatic infection, as well as to determine the percentage of personnel who have already passed the infection asymptomatically or to determine the percentage of personnel A healthcare provider who has developed some form of immunity following a confirmed COVID-19 infection.

The HUGTiP, like the rest of Catalan hospitals, has suffered a massive avalanche accumulated in the time of admission by COVID-19, which has forced it to adopt different innovative strategies to visit them in emergencies, enter them in conventional hospitalization in a conventional plant, or attend them in the intensive care units that had to be created de novo against the clock. As of April 20, 2020, 1,000 hospital discharges have been granted to patients admitted by COVID-19 in conventional hospitalization plants and 170 more discharges from those admitted to intensive care units at HUGTiP. Likewise, the Municipal Hospital of Badalona has given a total of 300 discharges of patients with COVID-19, and they have also reported about 180 infections in their health personnel in this period.

Due to the high transmission rate of SARS-CoV-2 and its potential severity, several healthcare workers at HUGTiP decided on their own to take empirical primary prophylaxis with oral hydroxychloroquine individually as prevention of SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age> 18 years) who have worked during the epidemic period (March and April 2020) in the Infectious Diseases, Pneumology, Emergencies, ICU and Internal Medicine departments of HUGTiP, or in the Internal Medicine or Emergency departments of the Badalona Municipal Hospital.

Exclusion Criteria:

* Participation will be voluntary and no exclusion criteria are established

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adults (age> 18 years) who have worked during the epidemic period (March and April 2020) in the Infectious Diseases, Pneumology, Emergencies, ICU and Internal Medicine departments of HUGTiP, or in the Internal Medicine or Emergency departments of the Badalona Municipal Hospital.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with past SARS-CoV-2 infection | Day 0
  Number of participants with past SARS-CoV-2 infection

SECONDARY OUTCOMES:
Number of infections in health personnel who have taken voluntary hydroxychloroquine as a prevention strategy for COVID-19 infection | Day 0
  Number of infections in health personnel who have taken voluntary hydroxychloroquine as a prevention strategy for COVID-19 infection
Number of infections in health personnel based on the degree of exposure to patients infected with COVID-19. | Day 0
  Number of infections in health personnel based on the degree of exposure to patients infected with COVID-19.
Number of infected participants who are active smokers and/or have chronic lung disease and/ or have history of hypertension.Relationship of degree of exposure to participants infected with SARS-CoV-2 admitted to the hospital.Professional category. | Day 0
  Number of infected participants who are active smokers and/or have chronic lung disease and/ or have history of hypertension.Relationship of degree of exposure to participants infected with SARS-CoV-2 admitted to the hospital.Professional category.
Number of participants infected with SARS-CoV-2 that presented symptoms and their grade. Number of participants infected with SARS-CoV-2 who required hospitalization. Number of participants infected with SARS-CoV-2 who received treatment. | Day 0
  Number of participants infected with SARS-CoV-2 that presented symptoms and their grade.
  Number of participants infected with SARS-CoV-2 who required hospitalization. Number of participants infected with SARS-CoV-2 who received treatment.
Number of family members infected from each participant with SARS-CoV-2 infection | Day 0
  Number of family members infected from each participant with SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Municipal de Badalona, Badalona, Barcelona